CLINICAL TRIAL: NCT05063318
Title: An Open-Label, Multicenter Study to Assess the Potential Effects of Itraconazole (a Strong CYP3A4 Inhibitor) on the Pharmacokinetics of Lurbinectedin (PM01183) in Patients With Advanced Solid Tumors
Brief Title: Clinical Trial of Lurbinectedin (PM01183) in Patients With Advanced Solid Tumors
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: PharmaMar (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: PM1183-A-018-20
Record Dates: First submitted 2021-09-02; First posted 2021-10-01 (Actual); Results first posted 2025-09-02 (Actual); Last update posted 2025-09-02 (Actual); Status verified 2025-08

CONDITIONS: Advanced Solid Tumors
MeSH Terms: interventions — PM 01183

STUDY DESIGN:
Intervention Model Description: This is a prospective, open-label, two-way crossover, phase Ib drug-drug interaction study in patients with advanced solid tumors.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Sequence TR (Active Comparator): Sequence 1 (TR)
  * Cycle 1: Itraconazole + lurbinectedin 0.8 mg/m²
  * Cycle 2: Lurbinectedin alone 3.2 mg/m²
  * Cycle 3: Lurbinectedin alone 3.2 mg/m² (optional)
  PART A The dose of lurbinectedin when given in combination with itraconazole for the initial three patients in Part A will be 0.8 mg/m². In Part A, all patients will receive itraconazole plus lurbinectedin in Cycle 1 and lurbinectedin alone in Cycles 2 and 3 (this last cycle being optional).
  PART B Randomization will apply for study Part B only. In Part B is susceptible to be adjusted properly if deemed necessary based on exposure and safety experience in Part A. In Part B, patients will be randomly assigned to the corresponding sequences.
  Interventions: Drug: Lurbinectedin alone; Drug: Lurbinectedin+Itraconazole co-administration
- Sequence RT (Active Comparator): Sequence 2 (RT):
  * Cycle 1: Lurbinectedin alone 3.2 mg/m²
  * Cycle 2: Itraconazole + lurbinectedin 0.8 mg/m²
  * Cycle 3: Lurbinectedin alone 3.2 mg/m² (optional)
  Interventions: Drug: Lurbinectedin alone; Drug: Lurbinectedin+Itraconazole co-administration

INTERVENTIONS:
Drug: Lurbinectedin alone — The dose of lurbinectedin during Parts A and B will be 3.2 mg/m² for all patients when administered without itraconazole.
Drug: Lurbinectedin+Itraconazole co-administration — The dose of lurbinectedin when given in combination with itraconazole for the initial three patients in Part A will be 0.8 mg/m², and in Part B is susceptible to be adjusted properly if deemed necessary based on exposure and safety experience in Part A.

SUMMARY:
Prospective, open-label, two-way crossover, phase Ib drug-drug interaction study in patients with advanced solid tumors

DETAILED DESCRIPTION:
Prospective, open-label, two-way crossover, phase Ib drug-drug interaction study in patients with advanced solid tumors.

The study will include a pre-treatment (screening) phase (within 14 days before the first lurbinectedin or itraconazole administration) followed by a treatment phase consisting of two lurbinectedin cycles, one cycle in combination with itraconazole and one cycle as single agent (in different order depending on the study sequence), and one additional third cycle of lurbinectedin as a single agent for patients who meet the continuation criteria and obtain a clinical benefit after the first two cycles, and then follow-up of adverse events if any.

ELIGIBILITY:
Inclusion Criteria:

1. Voluntary signed and dated written informed consent prior to any specific study procedure.
2. Male or female with age ≥ 18 years.
3. Eastern Cooperative Oncology Group (ECOG) performance status (PS) of ≤ 1 (App. 1).
4. Life expectancy > 3 months.
5. Pathologically confirmed diagnosis of advanced solid tumors [except for primary central nervous system (CNS) tumors], for which no standard therapy exists.
6. Recovery to grade ≤ 1 from drug-related adverse events (AEs) of previous treatments, excluding alopecia and grade 1/2 asthenia or fatigue, according to the National Cancer Institute Common Terminology Criteria for Adverse Events (NCICTCAE v.5).
7. Laboratory values within fourteen days prior to Day 1 of Cycle 1
8. Left ventricular ejection fraction (LVEF) by echocardiography (ECHO) or multiple-gated acquisition (MUGA) within normal range (according to institutional standards).
9. Evidence of non-childbearing status for women of childbearing potential (WOCBP). WOCBP must agree to use a highly effective contraceptive measure up to six months after treatment discontinuation. Valid methods to determine the childbearing potential, adequate contraception and requirements for WOCBP partners are described in App. 2. Fertile male patients with WOCBP partners should use condoms during treatment and for four months following the last investigational medicinal product (IMP) dose.

Exclusion Criteria:

1. Concomitant diseases/conditions:

   1. History or presence of unstable angina, myocardial infarction, congestive heart failure, or clinically significant valvular disease within last year.
   2. Symptomatic arrhythmia or any uncontrolled arrhythmia requiring ongoing treatment.
   3. Known cirrhosis, alcohol induced steatosis, or chronic active hepatitis. For hepatitis B, this includes positive test for both Hepatitis B surface antigen (HBsAg) and quantitative Hepatitis B polymerase chain reaction (PCR or HVB-DNA+). For hepatitis C, this includes positive test for both Hepatitis C antibody and quantitative Hepatitis C by PCR (or HVC-RNA+).
   4. History of obstructive cholestatic liver disease (suitable for stenting procedure) or biliary sepsis in the past 2 months.
   5. Known of active COVID-19 disease (this includes positive test for SARS-CoV- 2 in nasopharyngeal/oropharyngeal swabs or nasal swabs by PCR).
2. Symptomatic, progressive or corticosteroids-requiring documented brain metastases or leptomeningeal disease involvement. Patients with asymptomatic documented stable brain metastases not requiring corticosteroids during the last four weeks are allowed.
3. Use of (strong or moderate) inhibitors or inducers of CYP3A4 activity within three weeks prior to Day 1 of Cycle 1.
4. Use of CYP3A4 substrates such as HMG-CoA reductase inhibitors such as atorvastatin, lovastatin and simvastatin for which concomitant administration with strong CYP3A4 inhibitor is contraindicated (App 3).
5. Treatment with any investigational product within the 30 days before Day 1 of Cycle 1.
6. Women who are pregnant or breast feeding and fertile patients (men and women) who are not using an effective method of contraception (see App 2).
7. Psychiatric illness/social situations that would limit compliance with study requirements.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 14 (Actual)
Dates: Start 2020-10-07 (Actual); Primary Completion 2022-04-21 (Actual); Study Completion 2022-04-21 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Sara Martínez Gonzalez, MD, Study Director — PharmaMar; Rubin Lubomirov, MD, PhD, Study Director — PharmaMar
Locations (2):
- Spain (2):
  - Fundacion Jimenez Diaz, Madrid
  - Hospital HM Sanchinarro, Madrid

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 14 patients were included and treated at 2 sites: 3 in Part A in Sequence 1 (S1 TR: ITZ+lurbinectedin in Cycle 1) and 11 in Part B, of them 5 in S1 and 6 in Sequence 2 (S2 RT: ITZ+lurbinectedin in Cycle 2). In Part A, all patients were assigned to S1 TR, while in Part B, patients were randomly assigned at a 1:1 ratio to S1 TR or S2 RT.
  Patients participated between 7Oct2020 and 3Mar2022 (last follow-up). The 1st dose of the 1st cycle on 15Oct2020. The last dose of the last cycle on 7Feb2022.
Groups:
- Part A - S1 (TR): PART A The dose of lurbinectedin when given in combination with itraconazole for the initial three patients in Part A will be 0.8 mg/m². In Part A, all patients will receive itraconazole plus lurbinectedin in Cycle 1 and lurbinectedin alone in Cycles 2 and 3 (this last cycle being optional).
  Sequence 1 (TR)
  * Cycle 1: Itraconazole + lurbinectedin 0.8 mg/m²
  * Cycle 2: Lurbinectedin alone 3.2 mg/m²
  * Cycle 3: Lurbinectedin alone 3.2 mg/m² (optional)
  Lurbinectedin alone: The dose of lurbinectedin during Parts A and B will be 3.2 mg/m² for all patients when administered without itraconazole.
  Lurbinectedin+Itraconazole co-administration: The dose of lurbinectedin when given in combination with itraconazole for the initial three patients in Part A will be 0.8 mg/m², and in Part B is susceptible to be adjusted properly if deemed necessary based on exposure and safety experience in Part A
- Part B - S1 (TR): PART B Randomization will apply for study Part B only. In Part B is susceptible to be adjusted properly if deemed necessary based on exposure and safety experience in Part A. In Part B, patients will be randomly assigned to the corresponding sequences.
  Sequence 1 (TR)
  * Cycle 1: Itraconazole + lurbinectedin 0.8 mg/m²
  * Cycle 2: Lurbinectedin alone 3.2 mg/m²
  * Cycle 3: Lurbinectedin alone 3.2 mg/m² (optional)
  Lurbinectedin alone: The dose of lurbinectedin during Parts A and B will be 3.2 mg/m² for all patients when administered without itraconazole.
  Lurbinectedin+Itraconazole co-administration: The dose of lurbinectedin when given in combination with itraconazole for the initial three patients in Part A will be 0.8 mg/m², and in Part B is susceptible to be adjusted properly if deemed necessary based on exposure and safety experience in Part A
- Part B - S2 (RT): PART B Randomization will apply for study Part B only. In Part B is susceptible to be adjusted properly if deemed necessary based on exposure and safety experience in Part A. In Part B, patients will be randomly assigned to the corresponding sequences.
  Sequence 2 (RT):
  * Cycle 1: Lurbinectedin alone 3.2 mg/m²
  * Cycle 2: Itraconazole + lurbinectedin 0.8 mg/m²
  * Cycle 3: Lurbinectedin alone 3.2 mg/m² (optional) Lurbinectedin alone: The dose of lurbinectedin during Parts A and B will be 3.2 mg/m² for all patients when administered without itraconazole.
  Lurbinectedin+Itraconazole co-administration: The dose of lurbinectedin when given in combination with itraconazole for the initial three patients in Part A will be 0.8 mg/m², and in Part B is susceptible to be adjusted properly if deemed necessary based on exposure and safety experience in Part A.
Period: Overall Study
Arm/Group | Part A - S1 (TR) | Part B - S1 (TR) | Part B - S2 (RT)
Started | 3 | 5 | 6
Completed | 0 | 0 | 0
Not Completed | 3 | 5 | 6
Not completed — Progressive disease | 2 | 0 | 3
Not completed — Compassionate use | 1 | 3 | 3
Not completed — Adverse Event | 0 | 1 | 0
Not completed — Withdrawal by Subject | 0 | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Part A - S1 (TR) | Part B - S1 (TR) | Part B - S2 (RT) | Total
Number analyzed (Participants) | 3 | 5 | 6 | 14
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0
  Between 18 and 65 years | 1 | 3 | 4 | 8
  >=65 years | 2 | 2 | 2 | 6
Age, Continuous [Median (Full Range); unit: years] | 69 [49 to 72] | 64 [56 to 70] | 62 [56 to 72] | 63 [49 to 72]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3 | 2 | 4 | 9
  Male | 0 | 3 | 2 | 5
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White | 3 | 5 | 6 | 14
Region of Enrollment [Number; unit: participants]
  Spain | 3 | 5 | 6 | 14
ECOG PS [Count of Participants; unit: Participants] — Eastern Cooperative Oncology Group (ECOG) performance status (PS) The ECOG PS scale indicates increasing levels of disability, with 0 indicating fully active; 1, restricted in strenuous activity; 2, restricted in work activity but ambulatory and capable of self-care; 3, capable of limited self-care; 4, completely disabled; and 5, dead
  Participants
    0 | 1 | 4 | 5 | 10
    1 | 2 | 1 | 1 | 4
Weight [Median (Full Range); unit: kg] | 58.9 [49.9 to 73.9] | 66.6 [50.0 to 102.9] | 69.5 [62.8 to 90.5] | 67.5 [49.9 to 102.9]
Height [Median (Full Range); unit: cm] | 165 [159 to 171] | 163 [152 to 172] | 166.5 [153 to 182] | 165 [152 to 182]
Stage at diagnosis [Count of Participants; unit: Participants] — Stage measures how far a cancer has spread from its origin. The staging system used by CDC's National Program of Cancer Registries and the National Cancer Institute's Surveillance, Epidemiology, and End Results program is called Summary Stage.
  Participants
    Early | 1 | 1 | 2 | 4
    Locally advanced | 0 | 1 | 2 | 3
    Metastatic | 2 | 3 | 2 | 7
Primary tumor [Count of Participants; unit: Participants]
  Ovarian carcinoma | 1 | 0 | 3 | 4
  Lung | 0 | 1 | 2 | 3
  Endometrial carcinoma | 0 | 2 | 0 | 2
  Colon adenocarcinoma | 0 | 1 | 0 | 1
  Epidermoid carcinoma | 0 | 1 | 0 | 1
  Leiomyosarcoma | 0 | 0 | 1 | 1
  Mesothelioma | 1 | 0 | 0 | 1
  Pancreatobiliary adenocarcinoma | 1 | 0 | 0 | 1
Number of sites at baseline [Median (Full Range); unit: sites] | 4 [2 to 4] | 3 [2 to 5] | 2 [1 to 5] | 3 [1 to 5]
Sites at baseline [Count of Participants; unit: Participants]
  1 | 0 | 0 | 2 | 2
  2 | 1 | 2 | 2 | 5
  3 | 0 | 1 | 1 | 2
  >4 | 2 | 2 | 1 | 5
Time from diagnosis to first infusion [Median (Full Range); unit: years] | 2.6 [1 to 3.4] | 3.4 [2 to 13.8] | 3.5 [2.5 to 6.8] | 3.4 [1 to 13.8]
Prior surgery [Count of Participants; unit: Participants] — Prior surgery yes
  Participants | 2 | 3 | 4 | 9
Prior radiotherapy [Count of Participants; unit: Participants] — Prior radiotherapy yes
  Participants | 1 | 2 | 3 | 6
Number of prior lines [Median (Full Range); unit: lines] | 4 [2 to 4] | 3 [3 to 7] | 6 [3 to 9] | 4 [2 to 9]
Prior lines [Count of Participants; unit: Participants]
  2 lines | 1 | 0 | 0 | 1
  3 lines | 0 | 3 | 1 | 4
  ≥4 lines | 2 | 2 | 5 | 9
Number of prior chemotherapy lines [Median (Full Range); unit: Lines of chemotherapy] | 2 [2 to 4] | 3 [2 to 6] | 5 [3 to 11] | 4 [2 to 11]
Prior chemotherapy lines [Count of Participants; unit: Participants]
  2 lines | 2 | 1 | 0 | 3
  3 lines | 0 | 2 | 1 | 3
  ≥4 lines | 1 | 2 | 5 | 8

OUTCOME MEASURES:

1. Primary Outcome: Pharmacokinetic Analysis: Dose-adjusted AUC(0-∞)
Description: The primary parameter of interest for the statistical analysis will be plasma dose adjusted AUC(0-∞)
Time Frame: Day 1, 2, 3, 5, 8, 11, 15, 22 (Cycle 1,2,3) (each cycle is 21 days)
Population: The pharmacokinetic analysis included data from only PK - evaluable patients from study Part B and the same study population was used to perform the statistical analysis in evaluating the ITZ - lurbinectedin drug-drug interaction. Part A was meant to ensure the adequacy of the dose of lurbinectedin (0.8 mg/m²) when given in combination with itraconazole, and patients (n=3) were not randomized for treatment sequence, so they were not included in the main analysis, as pre-specified in protocol.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: μg·h/L/mg
Groups:
- ITZ+LRB: The pharmacokinetic analysis included data from only PK - evaluable patients from study Part B and the same study population was used to perform the statistical analysis in evaluating the ITZ - lurbinectedin drug-drug interaction.
- LRB Alone: The pharmacokinetic analysis included data from only PK - evaluable patients from study Part B and the same study population was used to perform the statistical analysis in evaluating the lurbinectedin alone.
Arm/Group | ITZ+LRB | LRB Alone
Number analyzed (Participants) | 8 | 8
μg·h/L/mg | 288.55 (73.9) | 105.8 (77.37)
Statistical Analysis 1: Comparison: ITZ+LRB vs LRB Alone; Test type: Superiority; ANOVA; ANOVA mixed-effects model included treatment, period and sequence as fixed effects, and patient (sequence) as a random effect; Least-squares geometric mean ratio = 272.73, 90% CI 2-sided [213.22 to 348.86]

2. Secondary Outcome: Pharmacokinetic Analysis: Dose-normalized AUC(0-t)
Description: The dose-normalized area under the concentration-time curve (AUC) will be calculated using the linear-log trapezoidal rule with extrapolation to infinity.
Time Frame: Day 1, 2, 3, 5, 8, 11, 15, 22 (Cycle 1,2,3) (each cycle is 21 days)
Population: The pharmacokinetic analysis included data from only PK - evaluable patients from study Part B and the same study population was used to perform the statistical analysis in evaluating the ITZ - lurbinectedin drug-drug interaction
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: μg·h/L/mg
Arm/Group | ITZ+LRB | LRB Alone
Number analyzed (Participants) | 8 | 8
μg·h/L/mg | 244.77 (91.89) | 103.4 (78.85)
Statistical Analysis 1: Comparison: ITZ+LRB vs LRB Alone; Test type: Superiority; ANOVA; [statistical method as in outcome 1, analysis 1]; Least-squares geometric mean ratio = 236.73, 90% CI 2-sided [177.35 to 316.00]

3. Secondary Outcome: Pharmacokinetic Analysis: Dose-normalized Cmax
Description: The maximum dose-normalized plasma concentration (Cmax) will be obtained directly from the experimental data.
Time Frame: Day 1, 2, 3, 5, 8, 11, 15, 22 (Cycle 1,2,3) (each cycle is 21 days)
Population: as for outcome 2
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: μg/L/mg
Arm/Group | ITZ+LRB | LRB Alone
Number analyzed (Participants) | 8 | 8
μg/L/mg | 25.91 (53.15) | 22.43 (53.75)
Statistical Analysis 1: Comparison: ITZ+LRB vs LRB Alone; Test type: Superiority; ANOVA; [statistical method as in outcome 1, analysis 1]; least-squares geometric mean ratio. = 115.51, 90% CI 2-sided [100.07 to 133.33]

4. Secondary Outcome: Pharmacokinetic Analysis: T1/2
Description: Terminal half-life (T1/2) will be obtained from the terminal rate constant calculated by linear regression using at least 3 observations.
Time Frame: Day 1, 2, 3, 5, 8, 11, 15, 22 (Cycle 1,2,3) (each cycle is 21 days)
Population: as for outcome 2
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: hours
Arm/Group | ITZ+LRB | LRB Alone
Number analyzed (Participants) | 8 | 8
hours | 101.36 (61) | 46.59 (17.12)
Statistical Analysis 1: Comparison: ITZ+LRB vs LRB Alone; Test type: Superiority; ANOVA; ANOVA mixed-effects model included treatment, period and sequence (TR or RT) as fixed effects, and patient (sequence) as a random effect; Least-squares geometric mean ratio. = 217.57, 90% CI 2-sided [151.81 to 311.82]

5. Secondary Outcome: Pharmacokinetic Analysis: Total Body Clearance (CL)
Description: Total body clearance (CL), calculated by dividing the administered dose by the AUC with extrapolation to infinity.
Time Frame: Day 1, 2, 3, 5, 8, 11, 15, 22 (Cycle 1,2,3) (each cycle is 21 days)
Population: as for outcome 2
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: L/h
Arm/Group | ITZ+LRB | LRB Alone
Number analyzed (Participants) | 8 | 8
L/h | 3.47 (73.9) | 9.45 (77.37)
Statistical Analysis 1: Comparison: ITZ+LRB vs LRB Alone; Test type: Superiority; ANOVA; [statistical method as in outcome 1, analysis 1]; Least-squares geometric mean ratio = 36.67, 90% CI 2-sided [28.66 to 46.9]

6. Secondary Outcome: Pharmacokinetic Analysis: Volume of Distribution
Description: Volume of distribution (both at steady state and based on the terminal phase) (Vss and Vz, respectively): Vss is an estimate that equals mean residence time times total body clearance. Vz, calculated dividing the administered dose by the product of the AUC with extrapolation to infinity by the terminal rate constant
Time Frame: Day 1, 2, 3, 5, 8, 11, 15, 22 (Cycle 1,2,3) (each cycle is 21 days)
Population: as for outcome 2
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: L
Arm/Group | ITZ+LRB | LRB Alone
Number analyzed (Participants) | 8 | 8
L | 418.68 (111.45) | 419.14 (58.58)
Statistical Analysis 1: Comparison: ITZ+LRB vs LRB Alone; Test type: Superiority; ANOVA; [statistical method as in outcome 1, analysis 1]; Least-squares geometric mean ratio = 99.89, 90% CI 2-sided [65.76 to 151.74]

ADVERSE EVENTS:
Time Frame: Three 21-days cycles
Groups:
- ITZ+LRB Cycle: The dose of lurbinectedin when given in combination with itraconazole for the initial three patients in Part A was 0.8 mg/m², and in Part B was susceptible to be adjusted properly if deemed necessary based on exposure and safety experience in Part A. Patients treated in Part A were not evaluable for PK but were evaluable for safety. For that reason, this arm is reported in the safety section but not in the PK section.
- LRB Alone Cycle: The dose of lurbinectedin during Parts A and B will be 3.2 mg/m² for all patients when administered without itraconazole.
Arm/Group | ITZ+LRB Cycle | LRB Alone Cycle
All-Cause Mortality (participants affected / at risk) | 1/13 | 1/14
Serious Adverse Events (participants affected / at risk) | 4/13 | 5/14
Other Adverse Events (participants affected / at risk) | 12/13 | 13/14
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | ITZ+LRB Cycle (N=13) | LRB Alone Cycle (N=14)
Alanine aminotransferase increased (Investigations) | 1 (1) | 1 (1)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 (2) | 1 (2)
Small intestinal obstruction (Gastrointestinal disorders) | 1 (1) | 1 (1)
Rhabdomyolysis (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1)
Intestinal obstruction (Gastrointestinal disorders) | 1 (2) | 1 (2)
Deep vein thrombosis (Vascular disorders) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | ITZ+LRB Cycle (N=13) | LRB Alone Cycle (N=14)
Neutropenia (Blood and lymphatic system disorders) | 7 (13) | 7 (13)
Constipation (Gastrointestinal disorders) | 1 (1) | 1 (1)
Vomiting (Gastrointestinal disorders) | 4 (7) | 4 (7)
Fatigue (General disorders) | 4 (6) | 4 (6)
Bone pain (Musculoskeletal and connective tissue disorders) | 1 (2) | 1 (2)
Dysgeusia (Nervous system disorders) | 1 (1) | 1 (1)
Syncope (Nervous system disorders) | 1 (1) | 1 (1)
Cough (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1)
Anaemia (Blood and lymphatic system disorders) | 1 (1) | 1 (1)
Thrombocytopenia (Blood and lymphatic system disorders) | 1 (2) | 1 (2)
Abdominal pain (Gastrointestinal disorders) | 1 (1) | 1 (1)
Intestinal pseudo-obstruction (Gastrointestinal disorders) | 1 (1) | 1 (1)
Nausea (Gastrointestinal disorders) | 5 (10) | 5 (10)
Stomatitis (Gastrointestinal disorders) | 1 (1) | 1 (1)
Stoma site infection (Infections and infestations) | 1 (1) | 1 (1)
Decreased appetite (Metabolism and nutrition disorders) | 1 (1) | 1 (1)
Hypercalcaemia (Metabolism and nutrition disorders) | 1 (1) | 1 (1)
Back pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1)
Acute kidney injury (Renal and urinary disorders) | 1 (1) | 1 (1)
Diarrhoea (Gastrointestinal disorders) | 0 (0) | 1 (1)
Tumour pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 1 (1)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The only disclosure restriction on the PI is that the sponsor can review results communications prior to public release and can embargo communications regarding trial results for a period that is more than 60 days but less than or equal to 180 days from the time submitted to the sponsor for review.

DOCUMENTS (2):
  • Study Protocol (2021-03-18): https://cdn.clinicaltrials.gov/large-docs/18/NCT05063318/Prot_000.pdf
  • Statistical Analysis Plan (2022-05-27): https://cdn.clinicaltrials.gov/large-docs/18/NCT05063318/SAP_001.pdf